CLINICAL TRIAL: NCT00003326
Title: A Phase II Trial of Paclitaxel (TAXOL) Administered as a Weekly One Hour Infusion in Patients With Advanced Esophageal Cancer
Brief Title: Paclitaxel in Treating Patients With Metastatic, Recurrent, or Unresectable Cancer of the Esophagus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066278; THERADEX-B97-4250; BMS-TAX/MEN.04; MSKCC-98018; NYU-9801; NCI-V98-1414
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2001-04

CONDITIONS: Esophageal Cancer
Keywords: stage IV esophageal cancer; recurrent esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients with metastatic, recurrent, or unresectable cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate of paclitaxel administered as a weekly one hour infusion in patients with metastatic, locally recurrent, or unresectable squamous cell carcinoma and adenocarcinoma of the esophagus. II. Evaluate the safety of paclitaxel in this patient population. III. Assess the overall survival and quality of life of these patients.

OUTLINE: This is an open label, multicenter study. Patients receive intravenous paclitaxel over 1 hour weekly. Each course consists of four weeks. Patients receive treatment until disease progression or unacceptable toxic effects is observed. Patient response is assessed every 2 courses during the first year and then every 3 months in subsequent years. Quality of life is assessed prior to treatment, prior to each course for 6 courses, then every 2 courses. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic, locally recurrent, or unresectable squamous cell carcinoma or adenocarcinoma of the esophagus The bulk of the tumor must involve the esophagus or gastroesophageal (GE) junction (for tumors extending between the GE junction into the proximal stomach) Gastric cancers with only minor GE junction or distal esophagus involvement are not eligible Measurable or evaluable disease No prior treatment for metastatic disease No brain metastases No osseous metastases as only site of disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL AST or ALT no greater than 2 times upper limit of normal (ULN) Renal: Creatinine no greater than 2 times ULN Calcium no greater than 12 mg/dL Cardiovascular: No New York Heart Association class III/IV heart disease No myocardial infarction within 6 months of study No congestive heart failure No unstable angina No clinically significant pericardial effusion or arrhythmia Neurologic: No concurrent peripheral neuropathy greater than grade 1 Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active serious infection or medical illness No history of hypersensitivity to drugs containing Cremophor (teniposide, cyclosporine, or vitamin K) No invasive malignancies within 5 years, except: Curatively treated basal or squamous cell carcinoma of the skin Curatively treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy within 4 weeks of study No concurrent immunotherapy Chemotherapy: No more than 1 prior chemotherapy regimen or chemotherapy/radiation therapy given in a neoadjuvant or adjuvant setting No prior chemotherapy within 4 weeks of study No concurrent chemotherapy Endocrine therapy: No prior hormonal therapy within 4 weeks of study Concurrent megestrol (Megace) allowed No other concurrent hormonal therapy Radiotherapy: No prior radiotherapy within 4 weeks of study No prior radiation to greater than 30% of bone marrow No more than 1 prior chemotherapy/radiation therapy regimen given in a neoadjuvant or adjuvant setting No concurrent radiotherapy Surgery: No prior surgery within 2 weeks of study Other: No prior parenteral antibiotics within 1 week of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1997-09

CONTACTS AND LOCATIONS:
Overall Officials: David Paul Kelsen, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (30):
- United States (30):
  - Cancer Center of Southern Alabama, Mobile, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - Savannah Hematology Oncology Associates, Savannah, Georgia
  - Northwest Medical Specialists, P.C., Arlington Heights, Illinois
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Hospital, Worcester, Massachusetts
  - Missoula Medical Oncology P.C., Missoula, Montana
  - Nevada Cancer Center, Las Vegas, Nevada
  - University of Medicine and Dentistry of New Jersey - MOBILE, Newark, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Hollings Cancer Center, Charleston, South Carolina
  - Palmetto Hematology/Oncology Associates, Spartanburg, South Carolina
  - Harrington Cancer Center, Amarillo, Texas
  - Lone Star Oncology, Austin, Texas
  - Oncology Consultants, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin